CLINICAL TRIAL: NCT05700747
Title: Health Through Activity: A Pilot Study of a Rehabilitation Intervention for People Living With Multiple Myeloma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MGH Institute of Health Professions (Other)
Responsible Party: Principal Investigator, Kathleen Lyons, ScD, OTR/L, Principal Investigator, MGH Institute of Health Professions
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-437
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Results first posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Physical Therapy; Exercise Program
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health Through Activity (HTA) Intervention (Experimental): Participants will undergo study procedures as outlined:
  * Complete a baseline survey regarding activity level and quality of life.
  * Attend 6 weekly study visits at the MGH Institute of Health Professions IMPACT Practice Center.
  * Attend final study visit and complete the Satisfaction survey and an individual, semi-structured interview with site staff to supply feedback about the program.
  * After six weeks, complete the Satisfaction survey again.
  Interventions: Behavioral: Health Through Activity

INTERVENTIONS:
Behavioral: Health Through Activity — Six, weekly, customized sessions with licensed physical and occupational therapists.

SUMMARY:
The purpose of this study is to explore whether a structured program can help reduce the challenges of decreased physical functioning and quality of life for participants with multiple myeloma by providing a customized exercise program and fostering engagement in meaningful activities.

The name of the study intervention involved in this study is:

Health Through Activity (HTA) (six-session, rehabilitation exercise regimen)

DETAILED DESCRIPTION:
The goal of this single arm, pilot study of the Health Through Activity (HTA) rehabilitation intervention for people living with multiple myeloma is to determine if investigators can feasibly deliver the program out of the IMPACT Practice Center at the MGH Institute for Health Professions.

- The six-session 'Health Through Activity' program provides a customized exercise plan and encourages engagement in activities to reduce disability and improve quality of life.

* Study procedures including screening for eligibility, in-clinic visits, questionnaires, and surveys.
* Participation in this research study is expected to last up to 4 months.

It is expected that up to 20 people will take part in this research study.

An internal grant from the Massachusetts General Hospital Institute of Health Professions is providing equipment and staffing for this study.

ELIGIBILITY:
Inclusion Criteria:

-≥18 years of age

* Diagnosed with multiple myeloma currently receiving maintenance therapy,
* Experiencing disability as indicated by an answer of "yes" to the question "Do health problems interfere with your ability to carry out your social or day to day activities?"

Exclusion Criteria:

* Bone pain that is either a) new onset or increased in the past month or b) uncontrolled i.e., in the patient's estimation the bone pain "greatly interferes with daily activities"
* History of fracture in the past 12 months without fixation, or
* Any injury or medical condition that would prohibit being able to safely perform exercise as indicated by the Physical Activity Readiness Questionnaire[29] (i.e., atrial fibrillation, chest pain or angina, uncontrolled high blood pressure or hypertension, loss of balance due to dizziness in the past 12 months, or loss of consciousness in the past 12 months).
* We will also exclude individuals with moderate or worse cognitive impairment as indicated by a score of 3 or less on the Callahan six item cognitive screening tool.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Lyons, ScD, OTR/L, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 16 patients were approached 11/16 were formally screened 6/11 were not interested/eligible 5/11 were interested and eligible 5/5 interested/eligible patients enrolled
Period: Overall Study
Arm/Group | Health Through Activity (HTA) Intervention
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Health Through Activity (HTA) Intervention
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (4.7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Males | 3
  Females | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 5
  Ethnicity: Non-Hispanic/Latino | 5

OUTCOME MEASURES:

1. Primary Outcome: Rate of Participant Enrollment
Description: Number participants enrolled / Number screened positive & eligible. A rate of at least 75% will indicate feasibility.
Time Frame: At screening
Measure: Count of Participants; unit: Participants
Arm/Group | Health Through Activity (HTA) Intervention
Number analyzed (Participants) | 5
Participants | 5

2. Primary Outcome: Assessment Completion Rate
Description: Defined as the number of participants completing each of the three study assessments to number of participants enrolled. A completion rate of 85% will indicate feasibility.
Time Frame: Up to 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Health Through Activity (HTA) Intervention
Number analyzed (Participants) | 5
Participants | 5

3. Primary Outcome: Screening Rate
Description: Number patients screened/ Number patients identified as potentially eligible. Screening rate of at least 75% will indicate feasibility
Time Frame: Up to 4 months
Population: Our outcome of Screening Rate depends on a denominator of "Number patients identified as potentially eligible." Therefore, this number is larger than the 5 participants who enrolled/started the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Health Through Activity (HTA) Intervention
Number analyzed (Participants) | 16
Participants | 11

4. Primary Outcome: Eligibility Rate
Description: Number patients screening positive & eligible / Number screened. Eligibility rate is influenced by how many people in the clinical population are experiencing disability. Based on our pilot study, expected rate to be at least 35%.
Time Frame: Up to 4 months
Population: Our outcome of Eligibility Rate depends on a denominator of "Number screened." Therefore, this number is larger than the 5 participants who enrolled/started the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Health Through Activity (HTA) Intervention
Number analyzed (Participants) | 11
Participants | 5

5. Secondary Outcome: Intervention Completion Rate
Description: Defined as at least 75% of participants complete all six sessions of Health Through Activity (HTA) and if the mean number of sessions is greater than or equal to 4.
Time Frame: Up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Health Through Activity (HTA) Intervention
Number analyzed (Participants) | 5
Participants | 5

6. Secondary Outcome: Participant Satisfaction
Description: Assessed by the Satisfaction survey which is a 7-item survey that is rated on a 5-point Likert scale. Any item on the Satisfaction survey that generates a mean score of < 4 will trigger consideration of modification to the HTA program.
Time Frame: Up to 4 months
Population: 5/5 participants engaged in one-on-one semi-structured qualitative interviews following completion of intervention which allowed us to gauge overall participant experiences/satisfaction within the study and intervention. Unfortunately, a protocol deviation (reported to the IRB) resulted in the 7-item satisfaction survey not being included in the data collection materials. This measure will not be collected as participants had already completed the program and study will be closed to enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Health Through Activity (HTA) Intervention
Number analyzed (Participants) | 5
Participants
  Participants felt well supported by the interventionists | 5
  Participants described feeling connected to the interventionists. | 3
  Optimism and openness of interventionists kept participants engaged | 3
  Participants felt the program structure was both effective and adaptable to their needs | 5
  Participants identified areas of growth | 5
  The program catalyzed participants to stay engaged, take action, and reflect on progress | 5
  Suggestion to tailor messaging/advertising for better clarity of target audience. | 1
  Suggestion to highlight that the program can be adapted to various performance levels | 2
  Suggestion to explain why program addresses a wide range of health aspects vs going deep on one | 3

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up (up to 4 months)
Arm/Group | Health Through Activity (HTA) Intervention
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-06): https://cdn.clinicaltrials.gov/large-docs/47/NCT05700747/Prot_SAP_000.pdf